CLINICAL TRIAL: NCT05440474
Title: A Reliability and Validity Study of Urdu Version of COPENHAGEN Neck Functional Disability Scale in Patients With Chronic Neck Pain
Brief Title: Urdu Version of COPENHAGEN Neck Functional Disability Scale: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0287
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Disability Physical
Keywords: COPENHAGEN Neck Functional Disability Scale; Urdu Version; Reliability; Validity; Neck Disability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* The objective of the research is to do translation and to culturally familiarize the COPENHAGEN Neck Functional Disability Scale into the Urdu language.
* To investigate if the COPENHAGEN Neck Functional Disability Scale is reliable and validate in the Pakistani population with Chronic Neck pain.
* To check the correlation with Neck Disability Index, Neck Pain and Disability Scale.

DETAILED DESCRIPTION:
The English version of the COPENHAGEN Neck Functional Disability Scale will be translated into Urdu and culturally adapted, as per a previous recommendation. The COPENHAGEN Neck Functional Disability Scale will be given to participants who have consented, and would be chosen based on convenience sampling and inclusion and exclusion criteria. The inter-observer and intra-observer reliability of the COPENHAGEN Neck Functional Disability Scale, Neck Pain and Disability Scale , and Neck Disability Index will be evaluated in this study. On the same day, the questionnaire will be filled out created two times. An Inter - observer assessment will be done with 2 hour break between distributions of questionnaires. The initial observer then will gather a third assessment over one-week period. For data entry and analysis, Statistical Package of Social Sciences Version 23 will be utilized. Internal consistency will be checked using the Cronbach alpha value, and test retest reliability will be assessed using the Intra-class coefficient.

ELIGIBILITY:
Inclusion Criteria:

* From 20 years Old to 60 Years Old
* Participants with chronic Neck pain
* The patient having minimum cervical ROM and pain.
* Patient not taking medicine.
* No intervention between the test-retest assessments.

Exclusion Criteria:

To complete the forms because of a psychological Impairment, history or presence of;

* Rheumatic diseases, severe articulation inflammation, and cardiac disease.
* History of previous cervical or thoracic spine injury
* Any systematic disease with an unstable spine
* Illiteracy or lack of understanding of Urdu Language
* The presence of neurologic or musculoskeletal disorders other than the Neck Condition.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pakistani population with Chronic Neck pain will be part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
COPENHAGEN Neck Functional Disability Scale | day 1
  Item 1 & 5 on this three-dimensional scale assess pain severity, while items 2, 3, 4, 5, 7, 8, 9, 10, and 12 assess disability in everyday tasks, while items 6, 9, 11, 13, and 14 assess social contacts and recreational activities. The entire score varies from 0 to 30
Neck Pain and Disability Scale | day 1
  The Neck Pain and Disability Scale is a multidimensional form with 20 items that cover four dimensions: neck issues, pain intensity, the impact of neck pain on emotion, and the impact of neck pain on daily activities
Neck Disability Index | day 1
  Neck Disability Index includes ten questions that assess pain intensity, personal care, lifting, reading, headaches, attention, work, driving, sleeping, and recreational activities. Every question is graded on a scale of 0 to 5 (no disability to total disability).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No